CLINICAL TRIAL: NCT02839265
Title: FLT3 Ligand Immunotherapy and Stereotactic Radiotherapy for Advanced Non-small Cell Lung Cancer
Acronym: FLT3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-5267
Record Dates: First submitted 2016-07-15; First posted 2016-07-20 (Estimated); Results first posted 2024-06-06 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SBRT + FLT3 Ligand Immunotherapy (Experimental): Patients will be treated with stereotactic body radiotherapy (SBRT) to a single pulmonary or extrapulmonary lesion as well as FLT3 immunotherapy.
  FLT3 Ligand Therapy (CDX-301)
  * Daily subcutaneous injections of CDX-301 (75 ug/kg) will be administered for 5 days, beginning on the first day of SBRT.
  * Additional cycles of SBRT (to distinct lesions) and CDX-301 may be administered every 2-4 months to subjects who demonstrate evidence of clinical benefit (lack of treatment-related toxicity and no disease progression).
  * Study therapy will be discontinued in cases of treatment-related toxicity or disease progression.
  Interventions: Drug: FLT3 Ligand Therapy (CDX-301); Radiation: Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Drug: FLT3 Ligand Therapy (CDX-301) — See Arm 1 descriptions
Radiation: Stereotactic Body Radiotherapy (SBRT) — See Arm 1 descriptions
  Other Names: Stereotactic Ablative Radiotherapy (SABR)

SUMMARY:
Based on promising data from our laboratory demonstrating synergy between ablative local radiotherapy and FLT3 ligand immunotherapy in murine NSCLC models, investigators are performing a phase II study combining FLT3L immunotherapy and SBRT for patients with advanced NSCLC that has progressed following standard systemic therapy. All patients will receive daily subcutaneous injections of CDX-301 (75 µg/kg) for 5 days, beginning on the first day of SBRT. SBRT will be delivered to a single pulmonary or extrapulmonary lesion. The SBRT regimen will depend on the size and location of the target lesion. The primary endpoint will be progression-free survival at 4 months, defined using immune-related response criteria (irRC).

DETAILED DESCRIPTION:
Primary Objective

* To explore the efficacy of combining stereotactic body radiotherapy (SBRT) with FLT3 ligand immunotherapy for advanced non-small cell lung cancer (NSCLC).

Secondary Objectives

* To establish the feasibility and safety of combining SBRT with FLT3 ligand immunotherapy for advanced NSCLC.
* To quantify and evaluate potential surrogate outcomes for clinical efficacy of this treatment approach, including radiographic responses, immunologic responses, and circulating tumor cell levels.

ELIGIBILITY:
Inclusion Criteria:

* AJCC stage 3 or 4 histologically proven NSCLC not amenable to curative therapy
* Age >= 18 years
* Prior treatment with at least one standard chemotherapy regimen or targeted agent prior to enrollment
* Radiological assessment within 21 days prior to study entry demonstrating measurable disease that includes at least one pulmonary lesion . 1 cm in greatest dimension that would be amenable to SBRT and at least one measurable lesion that would be outside of the SBRT treatment fields
* History/physical examination within 30 days prior to registration
* ECOG performance status 0-2
* Signed, written informed consent

Exclusion Criteria:

* Less than 21 days between registration and the last receipt of chemotherapy, biotherapy, immunotherapy, radiotherapy (excluding palliative radiotherapy), or major surgery. Prior receipt of immunomodulatory therapy (eg: nivolumab) is permitted, as long as there has been a 21 day washout period following the most recent treatment.
* Untreated central nervous system metastases. Patients with a history of brain metastases must have had no CNS-directed therapy within the past 60 days and radiological assessment within 30 days of study entry demonstrating a lack of progressive CNS disease
* Ongoing or recent (within 21 days prior to study entry) use of high dose oral corticosteroids (.2 mg of dexamethasone daily or equivalent). Intranasal and/or inhaled corticosteroid use is permitted.
* Any unresolved CTCAE grade >2 toxicity from previous anti-cancer therapy. Patients with irreversible toxicity that is not reasonably expected to be exacerbated by study therapy (eg, hearing loss)may be enrolled after discussion with the principal investigators.
* History of allogeneic organ transplant or autoimmune disease
* Active malignancy, other than NSCLC, for which systemic therapy is indicated. History of adequately treated local basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer, asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy asides from hormonal therapy, adequately treated stage 1 or 2 cancer currently in complete remission, or any other cancer that has been in complete remission for >= 5 years is permitted.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements as judged by the treating physicians
* The following laboratory results, within 10 days of first study drug administration:

  * Hemoglobin . 9.0 g/dL, Absolute neutrophil count . 1.5 x 109/L, Platelet count . 100 x 109/L
  * Serum creatinine . 1.5 x ULN and creatinine clearance (by Cockcroft-Gault formula) < 60 mL/min
* Women of child bearing potential: positive pregnancy test (serum)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2024-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Ohri, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period spanned from July 2016 through 1/23/2020. All patients enrolled into the study were enrolled at Montefiore Medical Center.
Pre-assignment Details: 33 patients signed informed consent however 29 patients were enrolled and randomized into the study.
Groups:
- SBRT + FLT3 Ligand Immunotherapy: Patients will be treated with stereotactic body radiotherapy (SBRT) to a single pulmonary or extrapulmonary lesion as well as FLT3 immunotherapy.
  FLT3 Ligand Therapy (CDX-301)
  * Daily subcutaneous injections of CDX-301 (75 ug/kg) will be administered for 5 days, beginning on the first day of SBRT.
  * Additional cycles of SBRT (to distinct lesions) and CDX-301 may be administered every 2-4 months to subjects who demonstrate evidence of clinical benefit (lack of treatment-related toxicity and no disease progression).
  * Study therapy will be discontinued in cases of treatment-related toxicity or disease progression.
  FLT3 Ligand Therapy (CDX-301): See Arm 1 descriptions
  Stereotactic Body Radiotherapy (SBRT): See Arm 1 descriptions
Period: Overall Study
Arm/Group | SBRT + FLT3 Ligand Immunotherapy
Started | 33
Completed | 29
Not Completed | 4
Not completed — Screen Failure | 2
Not completed — Death | 1
Not completed — Progression of SVC syndrome prior to treatment initiation | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics provided for the 29 patients who consented and completed the study. As noted in the participant flow module, 2 other patients screen failed, 1 patient died prior to treatment initiation, and 1 patient was removed from study prior to treatment due to disease progression.
Arm/Group | SBRT + FLT3 Ligand Immunotherapy
Number analyzed (Participants) | 29
Age, Customized [Count of Participants; unit: Participants]
  <= 50 years | 3
  51-60 | 3
  61-70 | 9
  71-80 | 12
  >81 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black | 8
  Hispanic | 9
  White | 11
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: The primary endpoint is progression-free survival rate at four months (PFS4), defined as the rate estimate of the percentage of patients who are alive and progression-free at 16 weeks (~4 months) after initiation of study therapy.
Time Frame: 4 Months
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT + FLT3 Ligand Immunotherapy
Number analyzed (Participants) | 29
Participants | 14

2. Secondary Outcome: Dose Limiting Toxicities (DLTs)
Description: The number of participants with evidence of DLTs will be tabulated. For the purposes of this study, a DLT will be defined as any grade 3-5 treatment-emergent adverse event toxicity, scored using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, and occurring within 30 days after treatment with SBRT in combination with FLT3 ligand therapy (after the first treatment cycle). Asymptomatic laboratory abnormalities (eg: leukocytosis) that do not require intervention will not be counted as DLTs. For subjects who receive more than one "cycle" of SBRT and FLT3 ligand, only adverse events that occur after the first cycle will be scored as potential DLTs.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT + FLT3 Ligand Immunotherapy
Number analyzed (Participants) | 29
Participants | 4

3. Secondary Outcome: Radiographic Response Rate Based on Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Radiographic Response will be scored using RECIST V1.1 criteria based on 1st post-treatment imaging to quantify objective measures of change in tumor burden. RECIST uses a max of 10 target lesions per patient to determine when tumors in cancer patients improve, stay the same, or worsen during treatment. RECIST will be used to quantify the percentage of patients demonstrating Complete Response (CR), Partial Response (PR), Stable Disease (SD), Progressive Disease (PD), as follows:
  CR - resolution of all target lesions to background levels PR - at least 30% decrease in sum of diameters of target lesions (noting baseline diameters) SD - neither sufficient shrinkage to qualify for PR or sufficient increase to qualify for PD (noting smallest sum on study) PD - at least 20% increase in sum of diameters of target lesions (noting smallest sum on study); absolute increase of 5mm must be demonstrated; >=1 new lesion is considered PD If no CT/PET at a specific timepoint = "Not Evaluable"
Time Frame: Up to 27 months post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT + FLT3 Ligand Immunotherapy
Number analyzed (Participants) | 29
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 4
  Stable Disease (SD) | 8
  Progressive Disease (PD) | 17
  Not Evaluable (NE) | 0

4. Secondary Outcome: Radiographic Response Rate Based on PET Response Criteria in Solid Tumors (PERCIST)
Description: Radiographic Response will be scored using PERCIST criteria based on the first PET imaging done. PERCIST is a set of rules that define when tumors in cancer patients improve, stay the same, or worsen during treatment, based on imaging data. PERCIST criteria will be used to quantify the percentage of patients demonstrating Complete Metabolic Response (CMR), Partial Metabolic Response (PMR), Stable Metabolic Disease (SMD), Progressive Metabolic Disease (PMD), or Not Evaluable (NE) as follows:
  CMR - complete resolution of 18F-FDG uptake, disappearance of all target lesions to background levels, no new 18F-FDG lesions PMR - reduction of a minimum of 30% in target measurable tumor 18F-FDG SUL peak, no increase >30% in all lesions; no new lesions SMD - no CMR, PMR or PMD; no new lesions PMD - >30% increase in 18F-FDG peak; OR visible increase in extent of tumor uptake; OR new 18F-FDG lesions If CT/PET was not done at a specific timepoint, result will be considered "Not Evaluable"
Time Frame: Up to 27 months post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT + FLT3 Ligand Immunotherapy
Number analyzed (Participants) | 29
Participants
  Complete Metabolic Response (CMR) | 0
  Partial Metabolic Response (PMR) | 9
  Stable Metabolic Disease (SMD) | 9
  Progressive Metabolic Disease (PMD) | 11
  Not Evaluable | 0

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the percentage of patients alive at 5 years post-randomization. Data of subjects without a death record will be censored on the last known survival date.
Time Frame: From date of treatment to date of death, up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT + FLT3 Ligand Immunotherapy
Number analyzed (Participants) | 29
Participants | 3

ADVERSE EVENTS:
Time Frame: Patients were monitored for the onset of Adverse Events for 32 weeks following treatment. Patients were assessed for All-cause Mortality up to 5 years
Arm/Group | SBRT + FLT3 Ligand Immunotherapy
All-Cause Mortality (participants affected / at risk) | 26/29
Serious Adverse Events (participants affected / at risk) | 23/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SBRT + FLT3 Ligand Immunotherapy (N=29)
Vomiting (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 2 — Verbatim Terms: Abdominal Pain, Left Upper Quadrant Pain, Epigastric Pain
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Chest Pain (Cardiac disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 2 — Verbatim Terms: Sinus Tachycardia, Tachycardia
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1 — Signification hemoglobin drop to <6
Leukocytosis (Blood and lymphatic system disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4
Sepsis (Infections and infestations) | 2
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1
Cardiac Arrest (Cardiac disorders) | 3
Acute Kidney Injury (Renal and urinary disorders) | 1
Stroke (Nervous system disorders) | 1
Disease Progression (Respiratory, thoracic and mediastinal disorders) | 11 — NSCLC
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SBRT + FLT3 Ligand Immunotherapy (N=29)
Cough (Respiratory, thoracic and mediastinal disorders) | 17
Fatigue (General disorders) | 21 — Verbatim Terms: Fatigue, Weakness
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17 — Verbatim Terms: Dyspnea, Shortness of Breath, Dyspnea on Exertion
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 — Verbatim Term: Peripheral Neuropathy
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 5 — Verbatim Terms: Skin Blister, Dermatitis
Anorexia (Metabolism and nutrition disorders) | 10 — Verbatim Terms: Anorexia, Loss of Appetite, Decreased Appetite
Nausea (Gastrointestinal disorders) | 7
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 — Verbatim Terms: Pain in Extremity; Pain in Lower Extremity
Vomiting (Gastrointestinal disorders) | 5
Hypotension (Vascular disorders) | 1
Fever (General disorders) | 1
Pain (General disorders) | 1 — Described as 'general'
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 — Verbatim Term: Vitiligo/Halo Nevi
Dizziness (Nervous system disorders) | 2
Non-cardiac Chest Pain (Musculoskeletal and connective tissue disorders) | 4 — Verbatim Terms: Chest Pain, Flank Pain, Non-cardiac chest pain No documentation of cardiac related-chest pain
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 — Verbatim Term: Sensory Neuropathy
Esophagitis (Gastrointestinal disorders) | 2
Pain - Suprapubic (Renal and urinary disorders) | 1 — Verbatim Term: Pain Suprapubic Area
Edema Limbs (General disorders) | 3 — Verbatim Terms: Edema - lower extremity; Edema bilateral lower extremity to shins; Edema left leg; bilateral leg edema; Edema - left shoulder/armpit
Dysphagia (Gastrointestinal disorders) | 1
Laryngeal Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 — Verbatim Term: Cough with Hemoptysis
Constipation (Gastrointestinal disorders) | 4
Chills (General disorders) | 1
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 2 — Verbatim Terms: Chest Wall Discomfort. Left Chest Wall Pain
Abdominal Pain (Gastrointestinal disorders) | 1 — Verbatim Terms: Abdominal Pain, Left Upper Quadrant Pain, Epigastric Pain
Anxiety (Psychiatric disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Injection Site Reaction (General disorders) | 1 — At site of FLT3L injection
Dry Eye (Eye disorders) | 1
Blurred Vision (Eye disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 — Left-sided
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Flu Like Symptoms (General disorders) | 1
Pelvic Pain (Reproductive system and breast disorders) | 1 — Verbatim Term: Pain - left hip/pelvic. Corresponds to an iliac crest metastasis visualized on recent PET/CT scan
Weight Loss (Investigations) | 1
Paresthesia (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT02839265/Prot_SAP_000.pdf